CLINICAL TRIAL: NCT07357142
Title: JING SI HERBAL TEA Use as Adjuvant Treatment in Patients With Chronic Pelvic Pain Syndrome
Brief Title: Jing Si Herbal Tea as Adjuvant Treatment in Patients With Chronic Pelvic Pain Syndrome
Acronym: JSHT-CPPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Chun-Kai Hsu, Attending Physician, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-IRB062; TCMF-JCT 115-06 (Other Grant/Funding Number: Buddhist Tzu Chi Medical Foundation)
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pelvic Pain Syndrome (CPPS)
Keywords: Chronic Pelvic Pain Syndrome; CPPS; Jing Si Herbal Tea; Herbal Medicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The placebo is identical in appearance and packaging to the investigational product to maintain the blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jing Si Herbal Tea Group (Experimental): Participants in this group will receive Jing Si Herbal Tea as an adjuvant therapy. They are instructed to take the tea orally twice daily (BID) - one pack in the morning and one in the evening - for a duration of 12 months.
  Interventions: Dietary Supplement: Jing Si Herbal Tea
- Placebo Control Group (Placebo Comparator): Participants in this group will receive a matching placebo. They are instructed to take the placebo orally twice daily (BID) - one pack in the morning and one in the evening - for a duration of 12 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Jing Si Herbal Tea — Oral administration, 2 packs daily (one in the morning and one in the evening) for 12 months.
  Arms: Jing Si Herbal Tea Group
Other: Placebo — Oral administration of a matching placebo, 2 packs daily (one in the morning and one in the evening) for 12 months. The placebo is identical in appearance and packaging to the investigational product.
  Arms: Placebo Control Group

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy of Jing Si Herbal Tea as an adjuvant treatment for patients diagnosed with Chronic Pelvic Pain Syndrome (CPPS). The study aims to determine whether adding Jing Si Herbal Tea to standard care can improve clinical symptoms and quality of life in these patients.

DETAILED DESCRIPTION:
Background: Chronic Pelvic Pain Syndrome (CPPS) is a clinically complex condition characterized by persistent pain, often accompanied by lower urinary tract symptoms and other physiological or psychological impacts. Patients frequently lack a definitive, single etiology, necessitating a multimodal treatment approach. Current standard management often involves the combined use of antibiotics (for prevention and treatment of bacterial infections), anti-inflammatory drugs (for symptom control), and alpha-blockers (to improve voiding symptoms). However, these treatments are associated with known side effects, concerns regarding future antibiotic resistance, and suboptimal efficacy in many patients. While local electrical stimulation and acupuncture are viable alternatives, accessibility and convenience remain significant barriers for patients.

Study Rationale: This study aims to evaluate the combined use of "Jing Si Herbal Tea" (JSHT) with standard pharmacological treatment. The objective is to alleviate patient symptoms, improve quality of life, reduce medication usage, and decrease healthcare expenditures.

Intervention Mechanism: Jing Si Herbal Tea (JSHT) is a multi-herbal formula containing various bioactive compounds known for their anti-inflammatory and immunomodulatory properties. It is proposed as an adjuvant therapy to alleviate symptoms of CPPS. The anti-inflammatory mechanism of JSHT is attributed to its active ingredients, including ovatodiolide, glycyrrhizin, eupatilin, and rosmarinic acid. These compounds exert their effects by inhibiting the NF-κB signaling pathway, reducing the secretion of pro-inflammatory cytokines (such as TNF-α and IL-6), and decreasing oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients.
2. Diagnosed with Chronic Pelvic Pain Syndrome (CPPS) at the investigational site.
3. Currently receiving continuous follow-up and medical treatment.

Exclusion Criteria:

1. Female patients (Excluded because the standard treatment, alpha-blockers, is not approved or reimbursed by the National Health Insurance for this indication in women in Taiwan).
2. Duration of symptoms less than 3 months.
3. History of recurrent urinary tract infections.
4. Diagnosed with malignancy.
5. Hospitalization for other diseases within the past 3 months.
6. Unwilling to participate in the study.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) Total Score | Baseline, Month 1, Month 2, Month 3, Month 6, and Month 12
  The NIH-CPSI is a standardized 9-item questionnaire used to assess symptom severity in patients with CPPS across three domains: Pain, Urinary Symptoms, and Quality of Life. The total score ranges from 0 to 43, with higher scores indicating more severe symptoms. Severity is categorized as Mild (0-14), Moderate (15-29), and Severe (30-43).

SECONDARY OUTCOMES:
Change in Short Form 12 Health Survey (SF-12) Score | Baseline, Month 1, Month 2, Month 3, Month 6, and Month 12
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It produces two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Scores range from 0 to 100, with higher scores indicating better health-related quality of life.
Incidence of Adverse Events | Up to 12 months
  Number of participants with treatment-related adverse events or side effects to evaluate safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and confidentiality. The informed consent form signed by participants does not include provisions for the public release of individual-level data.